CLINICAL TRIAL: NCT01354249
Title: Effects of Preoperative Feeding With a Whey Protein Plus Carbohydrate Drink on the Acute Phase Response and Insulin Resistance.
Brief Title: Preoperative Feeding With a Whey Protein Plus Carbohydrate Drink on the Acute Phase Response and Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Mato Grosso (Other)
Responsible Party: Jose Eduardo de Aguilar-Nascimento, Federal University of Mato Grosso
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: fperrone
Record Dates: First submitted 2011-05-10; First posted 2011-05-16 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Acute Phase Response; Insulin Resistance
Keywords: preoperative fasting; insulin resistance; carbohydrates; whey protein; inflammatory response
MeSH Terms: conditions — Acute-Phase Reaction; Insulin Resistance | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- water (Placebo Comparator): Patients will receive water 3h before operation in the same volume of the study group
  Interventions: Dietary Supplement: whey protein plus carbohydrate drink
- whey protein plus carbohydrate (Experimental): The CHO-P group will receive 474 ml (evening drink) or 237 ml (3h prior to operation drink) of a solution containing 14% whey protein (100% lactoalbumin), 86% carbohydrates (45% hydrolyzed corn starch and 55% sucrose) and 0% lipids (Resource® Breeze - Nestlé, São Paulo, Brasil)
  Interventions: Dietary Supplement: whey protein plus carbohydrate drink

INTERVENTIONS:
Dietary Supplement: whey protein plus carbohydrate drink — The CHO-P group received 474 ml (evening drink) or 237 ml (3h prior to operation drink) of a solution containing 14% whey protein (100% lactoalbumin), 86% carbohydrates (45% hydrolyzed corn starch and 55% sucrose) and 0% lipids (Resource® Breeze - Nestlé, São Paulo, Brasil)
  Other Names: Resource® Breeze - Nestlé, São Paulo, Brasil

SUMMARY:
Prolonged fasting may increase the organic response to trauma. Carbohydrate-based drinks have been tested and they may reduce insulin resistance. No study so far has aimed to examine the possible benefits of whey protein drink in the composition of preoperative drinks.

DETAILED DESCRIPTION:
The patients will be randomized into two groups: the carbohydrate-protein group (CHO-P) and the control group (CO). The patients will reeive a specific drink to their group on the evening prior to surgery and three hours before the operation. The CHO-P group will receive 474 ml (evening drink) or 237 ml (3h prior to operation drink) of a solution containing 14% whey protein (100% lactoalbumin), 86% carbohydrates (45% hydrolyzed corn starch and 55% sucrose) and 0% lipids (Resource® Breeze - Nestlé, São Paulo, Brasil) and the CO group will receive the same volume of water.

Outcome measures On the day of the surgery and on the first postoperative day blood samples will be collected for glucose, insulin, triglycerides, albumin, pre-albumin, CRP, and α-1-acid glycoprotein (α-1-GA) assays. HOMA-IR will be calculated

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-65 years-old)
* Both sexes
* Candidates to elective moderate operations such as open cholecystectomy, laparoscopic cholecystectomy and unilateral repair of inguinal hernia).

Exclusion Criteria:

* Acute cholecystitis
* Diabetes mellitus
* Chronic kidney failure
* Chronic liver disease ot serum bilirubin greater than 2 mg/dL, body mass index (BMI) above 35Kg/m2
* American Anesthesiologists Association (ASA) score above 2
* Gastro-esophageal reflux
* Gastroparesis or intestinal obstruction
* Patients with any non-compliance with the study protocol, or who had associated operations, or presented significant intraoperative occurrences, or experienced prolonged operations (lasting more than 3 hours) were also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
insulin resistance | Homa-IR will be assessed in two time points: baseline (2-3 h before operatio) and 24h after operation
  Insulin resistance will be assessed by Homa-IR

SECONDARY OUTCOMES:
acute-phase response | Assays for the various acute-phase proteins will be done 2-3h before operation and 24 h after the operation
  Assays for albumin, pre-albumin, C reactive protein and α-1-acid glycoprotein

CONTACTS AND LOCATIONS:
Overall Officials: Jose Aguilar-Nascimento, D, PhD, Principal Investigator — Federal University of Mato Grosso
Locations (1):
- Hospital Julio Muller, Cuiabá, Mato Grosso, Brazil

REFERENCES:
- [Derived] Perrone F, da-Silva-Filho AC, Adorno IF, Anabuki NT, Leal FS, Colombo T, da Silva BD, Dock-Nascimento DB, Damiao A, de Aguilar-Nascimento JE. Effects of preoperative feeding with a whey protein plus carbohydrate drink on the acute phase response and insulin resistance. A randomized trial. Nutr J. 2011 Jun 13;10:66. doi: 10.1186/1475-2891-10-66. PMID 21668975
- See also: Projeto Acerto — http://www.projetoacerto.com.br